CLINICAL TRIAL: NCT03438981
Title: Impact op Capillary Leak and Hypoalbuminemia on PK/PD of Ceftriaxone in Critically Ill Patients With Overwhelming Pneumonia
Brief Title: Optimization of PK/PD Target Attainment for Ceftriaxone in Critically Ill Patients With Community-acquired Pneumonia.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Matthias Gijsen, PharmD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: ML8457
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pharmacokinetics; Critical Illness
Keywords: Pharmacokinetics; Ceftriaxone; critical illness; capillary leak; hypoalbuminemia
MeSH Terms: conditions — Critical Illness; Hypoalbuminemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Serum Urine Broncho-alveolar lavage fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
WP2.1. PK/PD target attainment Plasma exposure ELF exposure WP2.2. Predictive dosing algorithm WP2.3. ECMO subset

DETAILED DESCRIPTION:
First, the investigators will document exposure to ceftriaxone in plasma and epithelial lining fluid.

Second, the investigators will try to identify risk factors for not attaining PK/PD target. Based on significant predictors for target non attainment a predictive dosing algorithm will be constructed.

Finally in a small subset of ECMO patients PK exposure will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia
* Admitted to an ICU ward
* Treated with ceftriaxone

Exclusion Criteria:

* Pregnancy
* DNR code 2-3
* Renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients receiving ceftriaxone treatment for pneumonia.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Risk factors for target non attainment | on day of sampling
  risk factors will be assessed by comparing patients who attain target vs. those who don't

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PhD PharmD, Study Director — isabel.spriet@uzleuven.be
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
To be discussed